CLINICAL TRIAL: NCT00001518
Title: A Randomized Evaluation of the Effect of Routine Normal Saline Flush Versus Heparinized Saline Solution in Groshong and Groshong PICC Catheters
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 960053; 96-CC-0053
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-12

CONDITIONS: Catheters, Indwelling; Thrombosis
Keywords: Groshong Catheter; Heparinized Flush Solution; Intraluminal Clot; Urokinase; Venous Access Device; Withdrawal Occlusion
MeSH Terms: conditions — Thrombosis

SUMMARY:
The Groshong and Groshong PICC catheters are popular venous access devices because they are maintained with only weekly saline flushes. In a recent study, however, we found an apparent decrease in the rate of withdrawal occlusion in Groshong catheters flushed weekly with heparinized saline. However, a randomized trial is necessary to confirm this impression. In the current study as many as 66 patients will be randomized to each of two treatment arms. The Groshong catheters of one group will be flushed with saline only and the other group with heparinized saline. A comparison will be made between the frequency with which urokinase is used in the two groups to treat withdrawal occlusion during the first three months of catheterization. Groshong catheters using saline flushes will be compared to Groshong catheters using heparinized saline flushes and Groshong PICC catheters using saline flushes will be compared to Groshong PICC catheters using heparinized saline flushes. Data will be analyzed using Fisher's exact test.

DETAILED DESCRIPTION:
The Groshong and Groshong PICC catheters are popular venous access devices because they are maintained with only weekly saline flushes. In a recent study, however, we found an apparent decrease in the rate of withdrawal occlusion in Groshong catheters flushed weekly with heparinized saline. However, a randomized trial is necessary to confirm this impression. In the current study as many as 66 patients will be randomized to each of two treatment arms. The Groshong catheters of one group will be flushed with saline only and the other group with heparinized saline. A comparison will be made between the frequency with which urokinase is used in the two groups to treat withdrawal occlusion during the first three months of catheterization. Groshong catheters using saline flushes will be compared to Groshong catheters using heparinized saline flushes and Groshong PICC catheters using saline flushes will be compared to Groshong PICC catheters using heparinized saline flushes. Data will be analyzed using Fisher's exact test.

ELIGIBILITY:
Adult subjects enrolled in approved protocols of the NCI in the CC or under treatment at the National Naval Medical Center who are planned to have Groshong Catheters used as part of their cancer treatment.

No subjects with a history of allergy to heparin.

No abnormal PT or PTT.

No subjects on anticoagulant therapy.

No history of heparin induced thrombocytopenia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 132
Dates: Start 1996-01; Study Completion 2000-11

CONTACTS AND LOCATIONS:
Locations (1):
- Warren G. Magnuson Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Mayo DJ, Horne MK 3rd, Summers BL, Pearson DC, Helsabeck CB. The effects of heparin flush on patency of the Groshong catheter: a pilot study. Oncol Nurs Forum. 1996 Oct;23(9):1401-5. PMID 8899756